CLINICAL TRIAL: NCT02205580
Title: Comparison of Three Different Rates of Continuous Intravenous Sufentanil Infusion for Postoperative Pain Management Following Coblation Tonsillectomy or Adeno-tonsillectomy in Children
Brief Title: Continuous Intravenous Sufentanil Infusion for Postoperative Pain Management Following Tonsillectomy or Adeno-tonsillectomy in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jin Ni (Other)
Responsible Party: Sponsor-Investigator, Jin Ni, Department of Anesthesiology, Guangzhou Women and Children's Medical Center
Organization: Guangzhou Women and Children's Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZWCMC
Record Dates: First submitted 2014-07-26; First posted 2014-07-31 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Sleep Breathing Disorders; Tonsillitis; Adenoid Hypertrophy
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sufentanil infusion rate 0.02μg•kg-1•h-1 (Experimental): Sufentanil infusion rate 0.02μg•kg-1•h-1 lasted for 48 hours
  Interventions: Drug: continuous intravenous sufentanil 0.02μg•kg-1•h-1 infusion
- Sufentanil infusion rate 0.03μg•kg-1•h-1 (Experimental): Sufentanil infusion rate 0.03μg•kg-1•h-1 lasted for 48 hours
  Interventions: Drug: continuous intravenous sufentanil 0.03μg•kg-1•h-1 infusion
- Sufentanil infusion rate 0.04μg•kg-1•h-1 (Experimental): Sufentanil infusion rate 0.04μg•kg-1•h-1 lasted for 48 hours
  Interventions: Drug: continuous intravenous sufentanil 0.04μg•kg-1•h-1 infusion

INTERVENTIONS:
Drug: continuous intravenous sufentanil 0.02μg•kg-1•h-1 infusion
  Arms: Sufentanil infusion rate 0.02μg•kg-1•h-1
Drug: continuous intravenous sufentanil 0.03μg•kg-1•h-1 infusion
  Arms: Sufentanil infusion rate 0.03μg•kg-1•h-1
Drug: continuous intravenous sufentanil 0.04μg•kg-1•h-1 infusion
  Arms: Sufentanil infusion rate 0.04μg•kg-1•h-1

SUMMARY:
Postoperative pain following tonsillectomy or adeno-tonsillectomy in children is severe and sometimes last for days. Sufentanil is used by epidural route for postoperative analgesia in children. There are few reports about its use for postoperative analgesia by continuous intravenous infusion. Its complications include , hypoxia, sedation, pruritus ,nausea and/or vomiting.

The investigators design this protocol to test efficacy of analgesia of three different rates of continuous intravenous sufentanil infusion for postoperative pain management following coblation tonsillectomy or adeno-tonsillectomy in children. The investigators also compare incidence rate of complications for three groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I or II children aged 5-8 years undergoing coblation tonsillectomy or adeno-tonsillectomy as in-patient

Exclusion Criteria:

* Children with a history of adverse reaction to opioids, long-term use of opioid medications, and history of chronic pain.
* Psychiatric illness, kidney failure, hypotension, atrioventricular block, myasthenia gravis etc.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
objective pain score | up to 48 hours after operation

SECONDARY OUTCOMES:
incidence rate of hypoxia | 4h,8h,24h,48h after operation

OTHER OUTCOMES:
incidence rate of pruritus | 4h,8h,24h,48h after operation
incidence rate of nausea and/or vomiting | 4h,8h,24h,48h after operation
incidence rate of sedation | 4h,8h,24h,48h after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ni, M.D., Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China